CLINICAL TRIAL: NCT01820130
Title: Trial of Autonomic neuroModulation for trEatment of Chronic Heart Failure
Acronym: TAME-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: end of inclusion period without patient enrolled
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-12-047-FR-SC
Record Dates: First submitted 2013-02-22; First posted 2013-03-28 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spinal Cord Stimulation system therapy (Experimental): St Jude Medical EON mini rechargeable system
  Interventions: Device: St Jude Medical EON mini rechargeable system

INTERVENTIONS:
Device: St Jude Medical EON mini rechargeable system — implantation of Eon Mini Neurostimulation System (IPG Model 3788)
  Other Names: Eon Mini Neurostimulation System (IPG Model 3788)

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and efficacy of Spinal Cord Stimulation (SCS) in advanced heart failure (HF) patients with Implantable Cardioverter Defibrillator (ICD) but not indicated for Cardiac Resynchronization Therapy (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Patients has a Left Ventricular Ejection Fraction (LVEF) less than or equal to 35%
* Patient is in New York Heart Association (NYHA) Class III
* Patient has a QRS duration <120 ms (non-paced QRS, at the time of device Implant or protocol inclusion)
* Patient has had an ICD implanted for >90 days
* Patient is receiving stable and optimal medical therapy for HF (>90 days) as describe by "European Society of Cardiology 2012 recommendation for diagnosis and treatment of acute and chronic Heart Failure", except in case of contraindication or allergy
* Patient is able to provide written Informed Consent prior to any investigational related procedure

Exclusion Criteria:

* Patient currently has an implanted spinal cord stimulator or previously had an implanted spinal cord stimulator which is now explanted or has had previous spinal surgery that would interfere with implant of percutaneous SCS leads in the upper thoracic region
* Patient has polyneuropathy
* Patient requires short-wave diathermy, microwave diathermy or therapeutic ultrasound diathermy
* Patient is in NYHA class IV
* Patient has received a tissue / organ transplant or is expected to have a tissue / organ transplant within the next 180 days
* Patient has a cardiac resynchronization therapy (CRT) device, or LV Assist device or is expected to receive CRT, or left ventricular assist device (LVAD) within the next 180 days
* Patient has critical valvular heart disease that requires valve repair or replacement
* Patient has had a myocardial infarction (MI) or cardiac revascularization procedure (percutaneous coronary intervention or coronary artery bypass graft) within 90 days of enrollment
* Patient is on IV inotropic therapy
* Patient has active myocarditis or early postpartum cardiomyopathy
* Patient has taken any of the following drugs within 30 days of enrollment: systemic corticosteroids, cytostatic and immunosuppressive drug therapy (cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.), DNA depleting or cytotoxic drugs
* Patient is pregnant, or of childbearing potential and is not using adequate contraceptive methods, or nursing
* Patient with a bleeding tendency (INR >1.2 and platelet count <100 x109 per liter)
* Patient has a local infection at the ICD implant location or systemic infection
* Patient has renal insufficiency (creatinine >3.0 mg/dl)
* Patient with risk of allergy to SCS device component materials
* Patient having one of the following condition must be considered as non relevant for SCS implantation:

  1. / Patient with active stent
  2. / Patient having bare metal stent for less than 6 months
  3. / Patient presented with an acute coronary syndrome within the last 6 months
  4. / Patient with stent on the common
  5. / Patient with a history of stent thrombosis
  6. / Coronary Patient receiving double antiplatelet medication
* Patient is participating in another clinical study with an active treatment arm
* Patient is less than 18 years old
* Patient's life's expectancy is less than 1 year as assessed by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy Marker of Cardiac remodeling via Left Ventricular End Diastolic Volume (LVEDV) of Patient with advanced HF | baseline and 6 Months
  Evaluation of left ventricular end diastolic volume (LVEDV) as measured by cardiac echo between baseline and after 6 months of SCS therapy.
Efficacy Marker of patient symptom via NYHA class for patient with advanced HF | Baseline and 6 months
  Evaluation of NYHA class as marker of patient symptom between baseline and after 6 months of SCS therapy.
Efficacy Marker of patient symptom via 6 Minutes Hall Walk distance for patient with advanced HF | baseline to 6 months
  Evaluation of 6 Minutes Hall walk (6MHW) as marker of patient symptom between baseline and after 6 months of SCS therapy.

SECONDARY OUTCOMES:
Safety composite marker of SCS therapy for patient with HF and ICD device | baseline and 6 months
  Report of cardiovascular event, arrythmias, devices interaction, procedural and post-procedural events analyzed in a global composite way.
Additional efficacy markers of SCS therapy on patient symptom via Quality Of Life questionnaire | baseline to 6 months
  Endpoint measurements of patient-reported quality of life after 6 months of therapy.
Additional efficacy markers of SCS therapy on patient symptom via Maximal exercise test tolerance | baseline and 6 months
  Additional endpoint measurements include exercise tolerance between baseline and 6 months via cardiopulmonary test, including maximum level of exercise and heart rhythm.
Additional efficacy markers of SCS therapy on cardiac function via echocardiography | baseline and 6 months
  Additional endpoint measurements include standard echocardiography markers of LV structure and function including systolic and diastolic performance and cardiac dimensions as a marker of structural reverse remodeling

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Bordachar, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU, Pessac, France